CLINICAL TRIAL: NCT02038712
Title: fMRI and Ghlrein in Obesity and Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Obesity and Nutrition Research Center (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Dr. Allan Geliebter, Senior Scientist, New York Obesity and Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 06-164
Record Dates: First submitted 2014-01-10; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Obesity; Binge Eating Disorder
Keywords: Obesity; Binge eating disorder; fMRI; gut hormones
MeSH Terms: conditions — Obesity; Binge-Eating Disorder | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Binge eating disorder (BED) (Experimental): Blood samples, subjective appetite ratings and fMRI scan will be collected in subjects who meet the current criteria for binge eating disorder (BED) in the fed condition and fasted condition.
  Interventions: Dietary Supplement: Fed Condition; Dietary Supplement: Fasted condition; Procedure: Blood samples; Behavioral: Subjective appetite ratings; Procedure: fMRI scan
- Control (Experimental): Blood samples, subjective appetite ratings and fMRI scan will be collected in subjects who do not meet the current criteria for BED (Controls) in the fed condition and fasted condition.
  Interventions: Dietary Supplement: Fed Condition; Dietary Supplement: Fasted condition; Procedure: Blood samples; Behavioral: Subjective appetite ratings; Procedure: fMRI scan

INTERVENTIONS:
Dietary Supplement: Fed Condition — Subjects will consume a 600mL 600kcal liquid test meal
  Other Names: Boost (Novartis Nutrition)
Dietary Supplement: Fasted condition — Subjects will consume 600mL plain water.
Procedure: Blood samples — Blood samples will be collected at -15, 0, 10, 30, 60, 90, 120 min
Behavioral: Subjective appetite ratings — Appetite ratings will be collected at -15, 0, 10, 30, 60, 90, 120 min.
Procedure: fMRI scan — Blood Oxygen Dependent (BOLD) signal response to pictures and words of food and non-food items will be measured using functional magnetic resonance imaging (fMRI).

SUMMARY:
Binge Eating Disorder (BED) may be associated with he development of obesity. However, the pathogenesis of BED is currently unclear, thus making the development of treatment and prevention strategies for BED difficult. Differences in the mechanisms regulating food intake may go some way to reveal potential mechanisms for BED.The purpose of this study is to investigate the responses of key gut-derived hormones that are associated with the regulation of food intake and functional brain activity to food cues using fMRI in BED patients and weight matched controls.

DETAILED DESCRIPTION:
Participants will attend the laboratory on two separate occasions following an overnight fast. Following baseline measures they will be provided wither with a 600mL (600kcal) liquid meal (Fed condition) or a volume matched amount of plain water (Fasted condition) to consume within 15 min in a randomized crossover design. Blood samples will be collected for during the subsequent 120min to measure the glucose, insulin and gut hormone responses, and subjective appetite ratings will be collected. 1500mg of acetaminophen will be added to each of the test drinks so that the appearance in the blood can be used as a proxy measure of gastric emptying. Participants will then undergo a 45min brain scan to assess the responses to visual and auditory food cues.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI 30-50 kg/m2
* Weight stable (<5% change in body weight during past 3 months)
* Right handed

Exclusion Criteria:

* Smokers
* Regular use of medications
* Current or intended participation in a weight-loss program (diet or exercise)
* Females who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
fMRI responses to food cues | 45 min
  Blood oxygen dependent signal (BOLD) response in exposure to auditory and visual food cues will be measured during a fMRI scan and the difference between responses in the fed condition compared with those in the fasted condition.

SECONDARY OUTCOMES:
Gut hormone responses | 120 min
  Blood samples will be collected at -15, 0, 10, 30, 60, 90, 120 min following the ingestion of the liquid test meal and analyzed to determine the gut hormone responses.
Subjective appetite ratings | 120 min
  Subjective ratings of appetite will be collected using a visual analogue scale (VAS) at -15, 0, 10, 30, 60, 90, 120 min following the liquid test meal

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — New York Obesity Nutrition Research Center